CLINICAL TRIAL: NCT02301572
Title: Aggressive Onset Multiple Sclerosis: A Practical Definition and Study of Its Clinical Course
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 0711009544
Record Dates: First submitted 2014-08-04; First posted 2014-11-26 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aggressive onset MS: Two or more relapses in the preceding year and 2 or more gadolinium enhancing lesions on brain MRI scan or a significant T 2 lesion burden or One relapse if it results in sustained EDSS of 3.0 along with 2 or more gadolinium enhancing lesions or significant T2 lesion burden ( T2 lesion burden being determined by factoring the number of lesions, the size of the lesions and lesion location)

SUMMARY:
Chart review.

DETAILED DESCRIPTION:
A chart review will be completed on patients with multiple sclerosis to determine potential early characteristics that might be helpful in defining aggressive onset MS and predicting subsequent disease course and disability

ELIGIBILITY:
Inclusion Criteria:

* Two or more relapses in the preceding year and 2 or more gadolinium enhancing lesions on brain MRI scan or a significant T 2 lesion burden or
* One relapse if it results in sustained EDSS of 3.0 along with 2 or more gadolinium enhancing lesions or significant T2 lesion burden ( T2 lesion burden being determined by factoring the number of lesions, the size of the lesions and lesion location)

Exclusion Criteria:

-

Ages: 0 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MS.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Disability outcome will be determined based on EDDS. | at the last visit (average time frame from baseline to last follow up visit expected to be 36 months)
  Disability outcomes will be determined based on EDDS at last visit. EDSS at last follow up will be compared to EDSS at start of respective therapies and grouped into 3 categories: EDSS improved, EDSS no change and EDSS worsened. Multivariate logistic regression will be used to test individual variables that could potentially influence the outcome, including treatment, age at onset, gender and race.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Perumal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No